CLINICAL TRIAL: NCT00561171
Title: A Phase IIa, Double-Blind, Randomized, Parallel-Design, Four-Week Study to Investigate the Efficacy and Safety of Two Different Doses of the Renin-Inhibitor SPP635 Once Daily in Type II Diabetic Patients With Mild to Moderate Hypertension and Albuminuria
Brief Title: Phase IIa Study to Investigate the Efficacy and Safety of SPP635 in Diabetic and Hypertensive Patients With Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Speedel Pharma Ltd. (Industry)
Responsible Party: Rolf Schlosshauer / Expert Clinical Manager, Novartis Pharma AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPP635CRD05
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: Hypertension; Type II Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): high dose
  Interventions: Drug: SPP635
- 2 (Experimental): lower dose
  Interventions: Drug: SPP635

INTERVENTIONS:
Drug: SPP635 — oral once daily

SUMMARY:
This is a phase II a, double-blind, randomized, parallel-design, four-week study to investigate the efficacy, safety and tolerability of two different doses of SPP635 in type II diabetic patients with mild to moderate hypertension and albuminuria.

The total study duration for patients completing the entire study will be approximately 7 weeks including a 2 weeks Screening Phase, 1 week Wash-out Phase, 4 week Treatment Phase and 1 week Follow-up Phase.

All treatments other than certain antihypertensive drugs (which are to be washed-out) with an effect on BP and all antidiabetic treatments must be kept at stable dose during the whole study.

A maximum of 50 patients in total is planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* men or women, 18 to 75 years
* hypertension
* diabetes mellitus type II
* albuminuria

Exclusion Criteria:

* donation of blood in the past month
* significant illness
* history of malignancy
* Heart failure, stroke, myocardial infarction, transient ischaemic attack, or hypertensive encephalopathy within the past 6 months
* Current or past history of clinically significant electrocardiogram (ECG) abnormalities such as permanent 2nd degree atrioventricular (AV) block or higher, unstable angina, percutaneous transluminal coronary angioplasty (PTCA), coronary artery bypass graft (CABG) or cerebrovascular accident in the last three months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
ABPM | 28 days

SECONDARY OUTCOMES:
sitting PB | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Maria Nicolaides, Dr., Study Director — Speedel Pharma Ltd.
Locations (1):
- Dr. John Barton, Ballinasloe, Co Galway, Ireland